CLINICAL TRIAL: NCT00341796
Title: A Prospective Cohort Study of the Seroprevalence of, and Interventions to Decrease the Risk of Mother-to-Child Transmission of, Human Immunodeficiency Virus Type 1 (HIV) in Tamil Nadu, India
Brief Title: Interventions to Decrease the Risk of Mother-to-Child Transmission of HIV in India
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902214; 02-CH-N214
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-08

CONDITIONS: HIV-1
Keywords: AIDS; HIV; Perinatal; Transmission; Antiretroviral; Outcomes
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

SUMMARY:
This study, conducted in Tamil Nadu, India, was initiated in response to the developing epidemic of HIV/AIDS in India. It is divided into two stages, as follows:

Stage I

All women registered in the pregnancy clinics at the Namakkal District Hospital or the Rasipuram Government Hospital in the state of Tamil Nadu in India will be offered participation in an educational session on HIV infection and transmission. It will include a pre-educational assessment of knowledge, attitudes, and beliefs, and a post-educational assessment of knowledge about HIV infection and transmission. All women at the clinic, regardless of whether or not they participate in the educational and assessment sessions, will be offered HIV counseling and testing. The objectives of this stage of the study are to:

* Assess the acceptance of education about HIV infection and transmission among pregnant women at the participating sites and their knowledge, attitudes, and beliefs about HIV
* Assess the acceptance of voluntary counseling and HIV testing among pregnant women at these sites
* Determine the prevalence of infection among women who accept HIV testing at these sites

Stage II

Pregnant HIV-infected women at the pregnancy clinics at the Namakkal District Hospital or the Rasipuram Government Hospital who are 18 years of age or older will be offered enrollment in Stage II of this study. Participants will be followed during their pregnancy and until their baby is a year old. The baby will be a part of the study from birth to one year of age. After delivery, both the mother and baby will be followed with regularly scheduled visits that include a physical examination and blood test.

Treatment with the anti-AIDS drug zidovudine will be offered for both the mother and child. For the study protocol, the mother will receive the drug starting the 28th week of pregnancy and continuing through labor and delivery. The infants will start drug treatment within the first 24 hours of life and continue for 6 weeks. Women who do not choose to take zidovudine according to this schedule will be offered standard treatment with a shorter course of drug, beginning with the 36th week of pregnancy, and no preventative treatment for their infants. All women will be offered education and counseling about the risks and benefits of breastfeeding and the risk of HIV transmission through breastfeeding. The objectives of this stage of the study are to:

* Assess the safety and tolerability of zidovudine given according to this protocol
* Assess the acceptance of and adherence to the zidovudine regimen in the protocol
* Assess the acceptance of education and counseling about breastfeeding
* Determine the mother-to-child HIV transmission rates in this study
* Determine the rates of illness and death through 12 months after delivery
* Determine risk factors for mother-to-child transmission of HIV

DETAILED DESCRIPTION:
This study is divided into two stages. In Stage I, all women registered in the antenatal clinics at the Namakkal District Hospital or at the Rasipuram Government Hospital in the state of Tamil Nadu in India will be offered the opportunity to participate in an educational session on HIV infection and transmission. With informed consent, a systematic sample of the population will be asked to participate in a pre-educational session assessment of knowledge, attitudes, and beliefs, and in a post-educational assessment of knowledge, regarding HIV infection and transmission. All women will be offered voluntary HIV counseling and testing, irrespective of participation in the education session (those who refuse to participate although education offered) and in the pre- and post-educational assessments (those among the systematic sample who do not provide signed informed consent). The objectives of Stage I are: (1) to assess the acceptance of education regarding HIV infection and transmission among antenatal women at the participating clinical sites and, among a systematic sample of those offered such education, to assess knowledge, attitudes, and beliefs, as well as changes in knowledge; (2) to assess the acceptance of voluntary counseling and HIV testing among antenatal women at the participating clinical sites; and (3) to describe the HIV seroprevalence among antenatal women at the participating clinical sites who accept HIV testing. The main outcomes of interest are the proportions of women in the antenatal clinics who agree to undergo HIV testing and, of these, the proportion who are seropositive for HIV.

HIV seropositive women will be offered enrollment in Stage II (a prospective cohort study). All women enrolled in the prospective cohort study will be offered education and counseling regarding infant feeding, i.e. the risks and benefits of breastfeeding, factors which are likely to increase the risk of transmission through breastfeeding, and the potential advantages and disadvantages of early weaning from breastmilk and replacement feeding.

Women enrolled in the prospective cohort study at Rasipuram Government Hospital who meet eligibility criteria will be offered Protocol ZDV/NVP: zidovudine prophylaxis beginning at 28 weeks gestation (or as soon as possible thereafter up to 36 weeks gestation if late presentation for antenatal care or other reasons preclude initiation at 28 weeks) and continuing through labor until delivery, and one dose of nevirapine at the onset of labor or as soon as possible thereafter. Their infants will receive zidovudine beginning within the first 24 hours of life and continuing through the end of the sixth week of life, and one dose of nevirapine within 24 hours after birth. Those women who decline protocol ZDV/NVP, or who enroll after 32 weeks gestation, can receive the standard of care: the two dose nevirapine regimen. (Women enrolled at Namakkal District Hospital could receive the two-dose nevirapine regimen.)

The primary objectives of Stage II are: (1) to assess the safety and tolerability of protocol ZDV/NVP; (2) to assess the acceptance of, and adherence to, protocol ZDV/NVP; (3) to assess the acceptance of education and counseling regarding infant feeding; and (4) to describe the mother-to-child transmission rates, among HIV-infected women and their infants enrolled in the prospective cohort study. The secondary objectives of Stage II are: (1) to describe morbidity and mortality rates through 12 months after delivery/birth; and (2) to describe risk factors for mother-to-child transmission of HIV, among HIV-infected women and their infants enrolled in the prospective cohort study. The primary outcomes of interest are the safety and tolerability of protocol ZDV/NVP, the proportion of HIV-infected women who agree to receive protocol ZDV/NVP, the mother-to-child HIV transmission rate (overall as well as according to receipt of protocol ZDV/NVP and infant feeding modality), and risk factors for transmission.

ELIGIBILITY:
* INCLUSION CRITERIA:

Stage I:

Registration in the Antenatal Clinics, Namakkal District Hospital or Rasipuram Government Hospital.

Stage II:

Registration in the Antenatal Clinics, Namakkal District Hospital or Rasipuram Government Hospital.

Receipt of voluntary HIV counseling.

Signed informed consent for HIV testing.

Completion of HIV testing.

Confirmation of HIV infection (documented by ELISA and Western Blot reports) if rapid test result is positive.

Receipt of results of HIV testing.

Age 18 years or more.

Residence in Namakkal District, Tamil Nadu.

Confirmation of pregnancy based upon history (last menstrual period) and/or physical examination (documented by a physician's statement in the medical record) and/or ultrasound.

Willingness and intent to be followed at the antenatal clinic or by home visits for 1year after delivery.

Signed informed consent by the HIV-infected woman for maternal and infant enrollment into prospective cohort study before onset of labor.

INCLUSION CRITERIA FOR MATERNAL Zidovudine ADMINISTRATION:

Enrollment in the prospective cohort study between 24 and 32 weeks.

Between 28 and 36 weeks gestation at initiation of protocol ZDV.

Signed informed consent by the father of the HIV-infected woman's unborn child.

Stated intention to deliver at Namakkal District Hospital or Rasipuram Government Hospital.

Laboratory criteria (ascertained within 30 days before initial dispensation of the drug).

Hematology-a) Hemoglobin concentration greater than or equal to 8 grams per deciliter.; b) Absolute neutrophil count greater than or equal to 1000 cells per cubic millimeter; c) Platelet count greater than or equal to 75,000 cells per cubic millimeter.

Serum chemistries - a) AST (SGOT) less than 92.5 Units per liter; b) ALT (SGPT) less than 100 Units per liter; c) Creatinine concentration less than 2.1 milligrams per deciliter.

Urinalysis - Urine protein less than 2+ by dipstick test.

INCLUSION CRITERIA FOR INFANT PROTOCOL ZDV ADMINISTRATION:

Mother enrolled in the prospective cohort study.

At least 36 weeks gestation.

Signed informed consent by the father.

Delivered at Namakkal District Hospital or Rasipuram Government Hospital.

EXCLUSION CRITERIA:

Stage II

Clinical - Diagnosis of pre-eclampsia.

Failure to meet all inclusion criteria.

EXCLUSION CRITERIA FOR INFANT PROTOCOL ZDV ADMINISTRATION:

Clinical - severe congenital malformations or other condition(s) not compatible with life; Documented or suspected serious infectious, cardiac, respiratory, or metabolic illness, or other immediate life threatening condition making the infant unable to tolerate oral medication beginning the first 24 hours of life.

Laboratory - Hemoglobin of less than 13 grams per deciliter.

Failure to meet all inclusion criteria.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2002-06; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Nduati R, John G, Mbori-Ngacha D, Richardson B, Overbaugh J, Mwatha A, Ndinya-Achola J, Bwayo J, Onyango FE, Hughes J, Kreiss J. Effect of breastfeeding and formula feeding on transmission of HIV-1: a randomized clinical trial. JAMA. 2000 Mar 1;283(9):1167-74. doi: 10.1001/jama.283.9.1167. PMID 10703779